CLINICAL TRIAL: NCT01399203
Title: Contrast Medium Volume and Contrast-induced Nephropathy After Percutaneous Coronary Intervention
Acronym: CONVIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Hainan People's Hospital (Other); Guangdong Medical College (Other)
Responsible Party: Ning Tan, MD, Guangdong Cardiovascular Institute,Guangdong General Hospital
Other Study IDs: 2009X41
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2010-01

CONDITIONS: Contrast Induced Nephropathy
Keywords: contrast-induced nephropathy; contrast medium; creatinine clearance; percutaneous coronary intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- percutaneous coronary intervention: The investigators reviewed all consecutive patients who were undergoing percutaneous coronary intervention

SUMMARY:
To investigate the predictive value of the contrast media volume to creatinine clearance (V/CrCl) ratio for the risk of contrast-induced nephropathy (CIN) (i.e., within 48-72 h) and to determine a relatively safe V/CrCl cut-off value to avoid CIN in patients following PCI

DETAILED DESCRIPTION:
contrast media volume to creatinine clearance (V/CrCl) ratios were obtained from consecutive consenting patients after unselective PCI. Receiver-operator characteristic (ROC) curves were used to identify the optimal sensitivity for the observed range of V/CrCl. The predictive value of V/CrCl for the risk of CIN was assessed using multivariate logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* patients who agreed to stay in the hospital for 2-3 days after percutaneous coronary intervention
* provided written informed consent
* Creatinine Clearance:15-60ml/min

Exclusion Criteria:

* pregnancy
* lactation
* intravascular administration of an contrast medium within the previous seven days
* treatment with metformin
* aminoglycosides
* N-acetylcysteine (NAC)
* nonsteroidal anti-inflammatory drugs within the previous 48 h
* intake of nephrotoxic drugs within the previous seven days
* history of serious reactions to contrast mediums
* severe concomitant disease
* renal transplantation , or end-stage renal disease necessitating dialysis patients who died during percutaneous coronary intervention

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators reviewed all consecutive patients who were undergoing percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-10 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Contrast-Induced Nephropathy | 48-72 h
  Contrast-Induced Nephropathy was defined as an increase in serum creatinine of more than 0.5 mg/dl from the baseline within 48-72 h of contrast exposure

SECONDARY OUTCOMES:
Major adverse clinical events | 1 year
  Major adverse clinical events: death, requiring renal replacement therapy, 2nd myocardial infarction,target revascularization,acute heart failure, mechanical ventilation,2nd angina,tachyarrhythmia,hypotension,intra-aortic balloon pump and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Yong Liu, MD, Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Ning Tan, Guangzhou, Guangdong, China